CLINICAL TRIAL: NCT04798534
Title: Facilitating the Decentralization of Methadone Maintenance Therapy Services Into Communities in Vietnam
Brief Title: Intervention to Facilitate MMT/HIV Service Decentralization in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Chunqing Lin, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R34DA04378; R34DA043783 (NIH)
Record Dates: First submitted 2021-03-04; First posted 2021-03-15 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Opioid-use Disorder
Keywords: Vietnam; Service Decentralization; Methadone maintenance therapy; HIV; Community health setting
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): CHW in the intervention arm will receive intervention through a combination of in-person training sessions and internet support. MMT patients in the intervention arm can use a specially designed online platform to communicate with their CHW.
  Interventions: Behavioral: Service decentralization facilitation intervention
- Control group (No Intervention): The control group CHW will perform business as usual. Both control group CHW and MMT patients do not have access to the online platform.

INTERVENTIONS:
Behavioral: Service decentralization facilitation intervention — The intervention CHW will participate in three 60-minute intervention weekly sessions. During the intervention, CHW will be provided with the knowledge and skills to serve their MMT patients. The intervention sessions will also focus on enhancing the current service decentralization workflow so that the CHW can work with both their peer providers and their patients more efficiently. Two-times booster sessions will be offered before the 3- and 6-month survey for continued skill building for problem-solving. In addition to the group sessions, the intervention arm CHW will be encouraged to use a specially designed online platform to review the current policy and scientific findings, review their patients' treatment status, communicate with other providers, and provide instant consulting to their MMT patients. The MMT patients in the intervention condition can use the online platform to communicate with their CHW and view education materials disseminated by their MMT providers or CHW.
  Arms: Intervention group

SUMMARY:
Vietnam is currently decentralizing its methadone maintenance therapy (MMT) dispensing network to its local commune health centers (CHC), which provides a window of opportunity to study decentralization of harm reduction and HIV-related healthcare services into community-based healthcare settings. Commune health workers (CHW) in Vietnam have widespread misconceptions about harm reduction and perceived significant challenges associated with treating people who use drugs. Intervention effort is needed to address these issues to ensure a smooth implementation of the decentralized service model. This study is to pilot testing an intervention with a primary focus on process optimization in six CHC-based MMT distribution sites with 30 CHW and 90 MMT patients. The six CHC in Thai Nguyen Province of Vietnam will be randomized to either an intervention condition or a control condition. The intervention will be executed through a combination of in-person training and mobile phone application utilization. The intervention outcomes on CHW and MMT clients will be evaluated at baseline, 3-, and 6-months.

DETAILED DESCRIPTION:
The intervention pilot will be conducted in six commune health center (CHC)-based methadone maintenance therapy (MMT) distribution sites in Thai Nguyen Province of Vietnam. Five commune health workers (CHW) and 15 MMT clients will be recruited from each of the CHC (total n = 30 CHW and 90 MMT clients). The six CHC will be matched into pairs based on the current number of CHW and MMT patient load; and within each pair, the two CHC will be randomized into either a control condition or an intervention condition. The intervention contents will include the promotion of streamlined procedure, skill training, problem solving, knowledge acquisition, networking and support, and information sharing. The intervention will be delivered through a combination of service provider in-person training and mobile phone application utilization. Provider-level outcomes (e.g., CHW's MMT/HIV service provision) and client-level outcomes (e.g., treatment progress) will be measured at baseline, 3-, and 6-month follow-ups.

ELIGIBILITY:
MMT patients (n=90):

Inclusion criteria:

* Age 18 or over
* Currently seeking MMT services in one of the participating commune health centers
* Voluntary informed consent

Exclusion criteria:

* Having psychosis or neurological damage, or cannot understand the study purposes as judged by the recruiter in consultation with a clinic supervisor.
* Inability to give informed consent

CHW (n=30):

Inclusion criteria:

* Age 18 or over
* Currently working in one of the participating commune health centers and have direct contact with MMT clients
* Providing informed consent

Exclusion criteria:

• Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
CHW's service provision for MMT providers | From baseline to 3-month
  This outcome will be evaluated using the change in CHW's self-reported number of hours in a typical week they spend on providing services for their MMT patients in the following areas: treatment adherence and retention, physical and mental health, employment status, family issues, STI/HIV risk reduction, and healthcare utilization.
CHW's service provision for MMT providers | From baseline to 6-month
  This outcome will be evaluated using the change in CHW's self-reported number of hours in a typical week they spend on providing services for their MMT patients in the following areas: treatment adherence and retention, physical and mental health, employment status, family issues, STI/HIV risk reduction, and healthcare utilization.
Patients' adherence to MMT | From baseline to 3-month
  This outcome will be measured using the change in the number of days the client received an MMT dosage divided by the total number of days during an observation period. Any occurrence of a special event (including termination of MMT, a positive urine test, and/or a dosage change) will be documented in detail.
Patients' adherence to MMT | From baseline to 6-month
  This outcome will be measured using the change in the number of days the client received an MMT dosage divided by the total number of days during an observation period. Any occurrence of a special event (including termination of MMT, a positive urine test, and/or a dosage change) will be documented in detail.

SECONDARY OUTCOMES:
Patients' level of satisfaction with community-based services | From baseline to 3-month
  This outcome will be measured using the change in the Verona Service Satisfaction Scale for Methadone Treatment (VSSS-MT; Range: 7-28; higher score indicates higher level of service satisfaction)
Patients' level of satisfaction with community-based services | From baseline to 6-month
  This outcome will be measured using the change in the Verona Service Satisfaction Scale for Methadone Treatment (VSSS-MT; Range: 7-28; higher score indicates higher level of service satisfaction)
Patients' service preference | From baseline to 3-month
  This outcome will be measured by change in patients' indicated preference between centralized healthcare agencies and CHC when they have a list of hypothetical health conditions (including mental health issues, infectious diseases, when seeking HIV testing and treatment, and STI treatment etc.)
Patients' service preference | From baseline to 6-month
  This outcome will be measured by the change in patients' indicated preference between centralized healthcare agencies and CHC when they have a list of hypothetical health conditions (including mental health issues, infectious diseases, when seeking HIV testing and treatment, and STI treatment etc.)
Patients' addiction and HIV-related service utilization | From baseline to 3-month
  This outcome will be measured by the change in the number of recorded service encounters with service providers during the last three months. Specifically, HIV/AIDS-related service utilization, including HIV testing and diagnosis will be documented at baseline and every follow-up point during the study period.
Patients' addiction and HIV-related service utilization | From baseline to 6-month
  This outcome will be measured by the change in the number of recorded service encounters with service providers during the last three months. Specifically, HIV/AIDS-related service utilization, including HIV testing and diagnosis will be documented at baseline and every follow-up point during the study period.
CHW's level of adherence to the working procedure | From baseline to 3-month
  This outcome will be measured using the change in score of an adapted version of Primary Care Behavioral Health Provider Adherence Questionnaire (PPAQ).The scale consists of three subscales to measure the CHW's favorable, acceptable, and prohibited clinical behaviors as specified in the revised protocol (range: 20-100; higher score indicates higher level of adherence to the working procedure).
CHW's level of adherence to the working procedure | From baseline to 6-month
  This outcome will be measured using the change in score of an adapted version of Primary Care Behavioral Health Provider Adherence Questionnaire (PPAQ).The scale consists of three subscales to measure the CHW's favorable, acceptable, and prohibited clinical behaviors as specified in the revised protocol (range: 20-100; higher score indicates higher level of adherence to the working procedure).
CHW's knowledge in harm reduction and HIV/AIDS will be assessed using a set of true-or-false questions based on the previously developed assessments | From baseline to 3-month
  This outcome will be measured using the change in CHW's service knowledge, assessed using a set of true-or-false questions based on the previously developed assessments (range 0-17; higher score indicates' better knowledge in harm reduction and HIV/AIDS).
CHW's knowledge in harm reduction and HIV/AIDS will be assessed using a set of true-or-false questions based on the previously developed assessments | From baseline to 6-month
  This outcome will be measured using the change in CHW's service knowledge, assessed using a set of true-or-false questions based on the previously developed assessments (range 0-17; higher score indicates' better knowledge in harm reduction and HIV/AIDS).
CHW's perceived challenges and administrative burdens in treating MMT patients | From baseline to 3-month
  This outcome will be measured using change in CHW's perceived challenge and administrative burdens in treating MMT patients, from recruitment, retention to provide referrals/consultations, using the Connecticut Primary Care Survey items (range: 13-52; higher score indicates higher level of perceived challenges and burdens).
CHW's perceived challenges and administrative burdens in treating MMT patients | From baseline to 6-month
  This outcome will be measured using change in CHW's perceived challenge and administrative burdens in treating MMT patients, from recruitment, retention to provide referrals/consultations, using the Connecticut Primary Care Survey items (range: 13-52; higher score indicates higher level of perceived challenges and burdens).
CHW's job satisfaction | From baseline to 3-month
  This outcome will be measured using change in CHW's level of satisfaction with various aspects of their career and specialty, including practice in addictive treatment, working hours, working environment, and income (Bellingham's Job Satisfaction Survey; range: 17-65; higher score indicates higher level of job satisfaction).
CHW's job satisfaction | From baseline to 6-month
  This outcome will be measured using change in CHW's level of satisfaction with various aspects of their career and specialty, including practice in addictive treatment, working hours, working environment, and income (Bellingham's Job Satisfaction Survey; range: 17-65; higher score indicates higher level of job satisfaction).
CHW's stigma associated with substance use | From baseline to 3-month
  This outcome will be measured using change in CHW's substance use stigma using Substance Abuse Attitudes Survey (SAAS; range: 7-35; higher score indicates higher level of stigmatizing attitude towards patients who use substances).
CHW's stigma associated with substance use | From baseline to 6-month
  This outcome will be measured using change in CHW's substance use stigma using Substance Abuse Attitudes Survey (SAAS; range: 7-35; higher score indicates higher level of stigmatizing attitude towards patients who use substances).
CHW's stigma associated with HIV | From baseline to 3-month
  This outcome will be measured using change in CHW's HIV stigma using adapted items of Substance Abuse Attitudes Survey (adapted SAAS; range: 7-35; higher score indicates higher level of stigmatizing attitude towards patients living with HIV).
CHW's stigma associated with HIV | From baseline to 6-month
  This outcome will be measured using change in CHW's HIV stigma using adapted items of Substance Abuse Attitudes Survey (adapted SAAS; range: 7-35; higher score indicates higher level of stigmatizing attitude towards patients living with HIV).

OTHER OUTCOMES:
MMT patients' mental health | From baseline to 3-month
  This outcome will be measured using the change in the Patient Health Questionnaire (PHQ-9), without the last item measuring suicidal ideation (range 0-24; higher score indicates worse mental health).
MMT patients' mental health | From baseline to 6-month
  This outcome will be measured using the change in the Patient Health Questionnaire (PHQ-9), without the last item measuring suicidal ideation (range 0-24; higher score indicates worse mental health).
MMT patients' heroin use | From baseline to 3-month
  This outcome will be measured using the change in patients' self-reported heroin use in the past 30 days (yes/no).
MMT patients' heroin use | From baseline to 6-month
  This outcome will be measured using the change in patients' self-reported heroin use in the past 30 days (yes/no).

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Hygiene and Epidemiology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
After all data are de-identified, cleaned, and validated, and main findings are published, the study team will make study data available upon request with the scientific community. Data sets will be made available to those who make a direct request to the PI and indicate the data will be used for the purposes of research. No identifiers will be included in these data sets. Depending on the request, data may be made available only in the form of codebooks and aggregated frequencies, to protect participant confidentiality. The names of the communes where data are collected may not be released beyond the immediate study team to further protect the privacy of participants.
Time Frame: Upon request